CLINICAL TRIAL: NCT03254550
Title: Expanding Options for HIV Prevention Through Pre-exposure Prophylaxis in Hhohho Region, Swaziland
Brief Title: PrEP Demonstration Study in Swaziland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinton Health Access Initiative Inc. (Other)
Collaborators: Ministry of Health, Swaziland (Other Government); Heidelberg University (Other); Mylan Laboratories (Industry); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Swazi PrEP study
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: HIV Negative People Identified at Substantial Risk for HIV Infection
Keywords: PrEP

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge randomized design (there was no option for stepped-wedge design in the drop-down menu) with two sequences (each consisting of three healthcare facilities) and three periods.
Masking Description: Healthcare facilities will not be informed as to when they are expected to start implementing the intervention (the PrEP Promotion Package) until two weeks prior to the start of the intervention phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control phase (No Intervention): This is the provision of PrEP without the use of the PrEP Promotion Package. PrEP promotion in the control phase consists of each clinic displaying posters that advertise PrEP, pamphlets, and palm cards that patients can take home from the clinic.
- Intervention phase (Experimental): This is the provision of PrEP as in the control phase plus the addition of five PrEP promotion components, which constitute the PrEP Promotion Package (PPP). These five additions are: 1) a PrEP promotion video to be played in the waiting room, 2) T-shirts advertising PrEP to be worn by healthcare workers, iii) a flipchart to support healthcare workers' PrEP counseling, iv) an informational booklet for clients to take home, and v) self-risk assessment forms to be displayed in the waiting room.
  Interventions: Other: PrEP Promotion Package

INTERVENTIONS:
Other: PrEP Promotion Package — A PrEP promotion package will be developed to test if this will change uptake, acceptance, retention and PrEP knowledge
  Arms: Intervention phase

SUMMARY:
This stepped-wedge cluster-randomized trial is embedded in an 18-month observational cohort study that has the aim to assess the operationalization of oral Pre-Exposure Prophylaxis (PrEP) in Swaziland as an additional HIV combination prevention method among individuals at high risk of HIV infection. The trial aims to determine the effect of a healthcare facility-based PrEP promotion package on the number of clients who take up PrEP.

DETAILED DESCRIPTION:
The study will assess who will be reached with an introduction to and an offer of PrEP - and who will take up PrEP - when PrEP becomes available through different delivery points in the public-sector health system, including outpatient department (OPD), antenatal care (ANC), postnatal care (PNC) , family planning (FP) , and following HIV counseling and testing (VCT).

In addition to PrEP reach and PrEP uptake, the study aims to establish PrEP retention and average costs per client, by different health systems delivery points and to assess the effectiveness of a feasible and low-cost PrEP Promotion Package (PPP). The exact composition of PPP will be informed by findings from in-depth- interviews with clients, providers, and PrEP stakeholders. The effect of the PPP on the monthly number of clients who are initiated on PrEP will be studied using a stepped-wedge cluster-randomized design. Specifically, the trial will have two sequences with three healthcare facilities in each sequence, and three periods. In the first period, all healthcare facilities will be in the control phase; in the second period three healthcare facilities will implement the PPP; and in the third period all six healthcare facilities will implement the PPP.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV negative by rapid antibody test following the National HIV testing services (HTS) algorithm on the day of PrEP initiation
* > 16 years of age
* Willing and able to provide written informed consent
* Identified at substantial risk of acquiring HIV infection
* No current or recent illness (within past month) consistent with acute HIV infection in combination with a preceding high risk exposure for HIV
* No contraindications to the use of Tenofovir(TDF)/Lamivudine (3TC)
* Ready to adhere to PrEP and willing to attend the follow up evaluations including repeat HIV testing and monitoring for side-effects

Exclusion Criteria:

* Younger than 16 years of age
* Currently having symptoms of acute HIV infection
* Suspicion of window period following a potential exposure to HIV
* Body weight < 40 kg
* Creatinine clearance <60 ml/min
* Using other nephrotoxic drugs (e.g. aminoglycosides)
* Not willing to come for follow up visits every 3 months which will include HIV testing and counselling and monitoring for side-effects.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Uptake | 18 months
  The monthly number of clients who was initiated on PrEP

SECONDARY OUTCOMES:
Risk assessment | 18 months
  The monthly number of clients who underwent a risk assessment for PrEP eligibility
Substantial risk | 18 months
  The monthly number of clients who was identified as being at a substantial risk of acquiring HIV
Acceptance conditional on risk | 18 months
  % of HIV-negative clients at substantial risk for HIV infection who accepted a PrEP offer
Linkage | 12 months
  The monthly number of clients who either took up PrEP or were linked to antiretroviral therapy
Retention at 6 months | 6 months
  % of clients taking PrEP who were retained at six months after PrEP initiation. Retention was defined as attending all follow-up visits during the first 180 days after PrEP initiation not more than seven days after the scheduled appointment.
HIV incidence | 18 month
  % of clients initiated on PrEP who seroconverted during the first six months after taking up PrEP.

CONTACTS AND LOCATIONS:
Overall Officials: Sindy Matse, MPH, Principal Investigator — Eswatini National AIDS Program
Locations (6):
- Eswatini (6):
  - Hhukwini Clinic, Hhukwini, Hhohho Region
  - Horo Clini, Horo, Hhohho Region
  - Ndvwabangeni Nazarene Clinic, Ndvwabangeni, Hhohho Region
  - Ndzingeni Nazarene Clinic, Ndzingeni, Hhohho Region
  - Nfontjeni Clinic, Nfontjeni, Hhohho Region
  - Siphocosini Clinic, Siphocosini, Hhohho Region

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03254550/SAP_000.pdf